CLINICAL TRIAL: NCT03951740
Title: Validation of Two Wrist-worn Devices for the Assessment of Energy Expenditure in Patients With Chronic Heart Failure and Coronary Artery Disease.
Brief Title: Validation of Two Wrist-worn Devices for the Assessment of Energy Expenditure in Cardiac Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maxima Medical Center (Other)
Responsible Party: Principal Investigator, H.Kemps, Cardiologist, Principal Investigator, Maxima Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: W17.062
Record Dates: First submitted 2019-05-06; First posted 2019-05-15 (Actual); Last update posted 2019-05-15 (Actual); Status verified 2019-05

CONDITIONS: Coronary Artery Disease; Heart Failure With Reduced Ejection Fraction
Keywords: Fitbit Charge 2; Mio Slice; Validation study; Energy expenditure
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: This is a single-center validation study with a comparative design. Accuracy and responsiveness of two wrist-worn activity trackers will be assessed. 39 patients (19 with coronary artery disease with preserved left ventricular ejection fraction and 19 with heart failure with reduced left ventricular ejection fraction) will be included.
Masking Description: Masking not applicable
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Group of cardiac patients (Experimental): All patients completed the study wearing two wrist-worn activity trackers and the Oxycon mobile as reference method during a laboratory activity protocol.
  Interventions: Device: Fitbit Charge 2; Device: Mio Slice; Device: Oxycon Mobile

INTERVENTIONS:
Device: Fitbit Charge 2 — Energy expenditure (kcal) assessed by this activity tracker will be compared with indirect calorimetry (Oxycon Mobile) during a laboratory activity protocol. Two groups will be assessed: patients with stable coronary artery disease (CAD) and patients with heart failure with reduced ejection fraction (HFrEF).
Device: Mio Slice — Energy expenditure (kcal) assessed by this activity tracker will be compared with indirect calorimetry (Oxycon Mobile) during a laboratory activity protocol. Two groups will be assessed: patients with stable coronary artery disease (CAD) and patients with heart failure with reduced ejection fraction (HFrEF).
Device: Oxycon Mobile — The Oxycon Mobile will be used as the reference method/golden standard to calculate energy expenditure (kcal). This device (consisting of a face mask and gas analyzer unit) will be worn during the entire laboratory activity protocol.
  Two groups will be assessed: patients with stable coronary artery disease (CAD) and patients with heart failure with reduced ejection fraction (HFrEF).

SUMMARY:
Improving physical activity is a core component of secondary prevention and cardiac (tele)rehabilitation. Commercially available activity trackers are frequently used to monitor and promote physical activity in cardiac patients. However studies on the validity of these devices in cardiac patients are scarce. The aim of this study is to determine the accuracy and responsiveness of two wrist-worn activity trackers, Fitbit Charge 2 (FC2) and Mio Slice (MS), for the assessment of energy expenditure (EE) in cardiac patients.

DETAILED DESCRIPTION:
Introduction

Improving physical activity is a core component of secondary prevention and cardiac (tele)rehabilitation. Commercially available activity trackers are frequently used to monitor and promote physical activity in cardiac patients. However studies on the validity of these devices in cardiac patients are scarce. The aim of this study is to determine the accuracy and responsiveness of two wrist-worn activity trackers, Fitbit Charge 2 (FC2) and Mio Slice (MS), for the assessment of energy expenditure (EE) in cardiac patients.

Methods

Eligible patients are recruited by their cardiologist in the outpatient cardiology clinic. If a patient is willing to participate, he/she visits the Máxima Medical Centre once, to perform the study measurements.

EE assessed by both activity trackers is compared with indirect calorimetry (Oxycon Mobile) during a laboratory activity protocol consisting of 14 low-to-moderate intensity activities. The duration of the activities varies between 1 to 5 minutes, while total duration of the protocol is 39 minutes (resting time excluded) Two groups are assessed: patients with stable coronary artery disease (CAD) and patients with heart failure with reduced ejection fraction (HFrEF).

Sample size calculation

To achieve 80% power to detect an intraclass correlation coefficient (ICC) of 0.75 (excellent agreement) under the alternative hypothesis that the ICC is 0.35 (poor agreement), a sample size of 19 subjects per study group (i.e. CAD and HFrEF) is calculated.

Statistical analysis

Accuracy of FC2 and MS will be assessed by calculating mean EE and mean differences in EE compared to the criterion measure (Oxycon Mobile). To identify if agreement is between reasonable limits one-sample T-tests will be performed using mean differences. In addition, Bland-Altman plots will be created to illustrate the level of agreement with mean bias and 95% upper and lower limits of agreement (LoA). Moreover ICC using two-way mixed models with absolute agreement will used. Responsiveness of FC2 and MS will be assessed by using a paired T-test during walking and cycling at different intensities. Significance level will be set at p<0.05 for all analyses.

ELIGIBILITY:
Inclusion criteria heart failure patients:

* Patients with heart failure with reduced ejection fraction (LVEF < 40%) due to ischemic or dilating cardiomyopathy
* New York Heart Association Class II to III
* Speaking Dutch language

Exclusion criteria heart failure patients:

* Hemodynamically significant valvular disease
* Atrial fibrillation
* Peripheral vascular, neurological and orthopaedic conditions impairing exercise capacity
* Severe psychological or cognitive impairments

Inclusion criteria patients with coronary artery disease

* Stable coronary artery disease regardless of intervention (PCI or CABG)
* Speaking Dutch language

Exclusion criteria patients with coronary artery disease

* Left ventricular ejection fraction < 50%
* Hemodynamically significant valvular disease
* Atrial fibrillation
* Peripheral vascular, neurological and orthopaedic conditions impairing exercise capacity
* Severe psychological and cognitive impairments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2017-10-11 (Actual); Primary Completion 2018-06-27 (Actual); Study Completion 2018-06-27 (Actual)

PRIMARY OUTCOMES:
Agreement | During a laboratory protocol consisting of 14 low-to-moderate intensity activities (39 minutes in total, resting time excluded)
  Energy expenditure (measured in kcal) will be extracted from both activity trackers for each separate activity of the protocol as well as for the total protocol.
  Breath-by-breath oxygen uptake (VO2) and carbon dioxide production (VCO2) will be measured during the entire length of the protocol using the Oxycon Mobile (reference method). By using the Weir equation, energy expenditure (kcal) will be calculated from VO2 and VCO2.
  Agreement of energy expenditure measurement is assessed by using mean differences in energy expenditure measured by the activity trackers versus the Oxycon Mobile and by calculating an intra-class correlation coefficient.

SECONDARY OUTCOMES:
Responsiveness | Cycling at three different intensities (3 minutes at each intensity) and treadmill walking at three different intensities (3 minutes at each intensity))
  Responsiveness (i.e. ability to detect within-patients changes of energy expenditure measurement over time) of the activity trackers will be calculated by using a paired T-test during walking and cycling at different intensities.

CONTACTS AND LOCATIONS:
Overall Officials: Hareld Kemps, MD, PhD, Principal Investigator — Maxima Medical Center
Locations (1):
- Máxima Medical Centre, Veldhoven, North Brabant, Netherlands

IPD SHARING:
Plan to Share IPD: No